CLINICAL TRIAL: NCT00154960
Title: Establishing Novel Detection Techniques for Various Genetic-Related Diseases by Applying DHPLC Platform.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9300005565
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2004-06

CONDITIONS: Spinal Muscular Atrophy; Neonatal Hyperbilirubinemia; Colon Cancer
Keywords: Spinal muscular atrophy (SMA); SMN1/SMN2 gene; denaturing high-performance liquid chromatography (DHPLC); multiplex PCR; gene dose; carrier test; screen; stool; microsatellite
MeSH Terms: conditions — Muscular Atrophy, Spinal; Hyperbilirubinemia, Neonatal; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
In this, here we want to present a new method for analysis variation in gene copy number for patients and carriers of SMA. This is a relative quantitation method and, therefore, relies on the inclusion of one or more internal control or reference sequences; quantitation of DNA is relative to this reference sequence of known copy number. A peak height from within a potentially duplicated or deleted target region is amplified simultaneously with a disomic reference region in a multiplex PCR system.

DETAILED DESCRIPTION:
Proximal spinal muscular atrophy is an autosomal recessive disorder with an overall incidence of 1 in 10000 live births and a carrier frequency of 1 in 50. This severe neuromuscular disease is characterized by a degeneration and loss of alpha motor neurons of the spinal cord anterior horn cells, which results in progressive symmetrical weakness, atrophy of the proximal voluntary muscles, and infant death. Here, we present a new, rapid, simple and high reliable method to detect the SMN1 deletion and to determine the copy number of the SMN1 and SMN2 by denaturing high-performance liquid chromatography (DHPLC). We demonstrate that this assay is able to accurately distinguish 2 gene copies from 4 gene copies and it can identify SMA carriers and normal populations by the accurate determination of SMN copy number.

Fecal DNA testing is a promising tool for colorectal cancer screening. Researchers have shown that DNA to be a good marker since it is stable in the stool; it shed continuously; and, through the use of amplification tests, it can be detected in minute amounts. Many DNA mutations associated with the process of colon cancer carcinogenesis have been characterized. K-ras oncogene, adenomatous polyposis coli (APC), p53, and microsatellite markers are examples of genes targeted as DNA markers in stool testing because they are critical to the control of colorectal cell growth. Early clinical studies have shown that multitarget DNA testing has a 71% to 91% sensitivity for detection of cancer and a 55% to 82% sensitivity for detecting adenoma 1cm or larger. We design this study, by using the automated DHPLC analysis and the microsatellite markers set already at first, to stepwisely set-up a high throughput but sensitive and specific screen method for colorectal cancer screen.

Neonatal hyperbilirubinemia is a common problem and is of concern not only to pediatricians but also to the parents of neonates. Two key enzymes, UDP-glucuronosyl transferase 1A1 and heme oxygenase-1 (HO-1), that involve bilirubin metabolism are highly noticed. First, UGT1A1 is the key enzyme for bilirubin conjugation and mutations of UGT1A1 cause the unconjugated hyperbilirubinemias known as Crigler-Najjar syndrome and Gilbert's syndrome. The high allele-frequency of Gly71Arg and promoter polymorphism in UGT1A1 gene was found to be responsible for neonatal hyperbilirubinemia without obvious cause. Second, HO-1 is a rate-limiting enzyme in the heme metabolism and allows for the degradation of heme to biliverdin. Recently, Maruo et al. demonstrated that (16/17) breastfed Japanese infants with apparent prolonged jaundice had at least one mutation of the UGT1A1. These data suggested that that defects of UGT1A1 may be an underlying cause of the prolonged unconjugated hyperbilirubinemia associated with breast milk. However, to date the association between breastfed infants with severe hyperbilirubinemia and UGT1A1 gene mutation is still unclear. In this study, we will analyze the UGT1A1 and HO-1 genes of infants with unconjugated hyperbilirubinemia associated with breast milk to ascertain whether genetic factors are involved.

This project will contribute to apply DHPLC on establishing various novels, fast, and reliable applications for diagnosis of SMA and carrier detection of SMN1 and SMN2 genes, sensitive and specific screen method for colorectal cancer screen, and analyze the UGT1A1 and HO-1 genes of infants with unconjugated hyperbilirubinemia associated with breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Spinal muscular atrophy (SMA)

Exclusion Criteria:

* nil

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ning Su, MD,PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- Dept of Medical Genetics;National Taiwan University Hospital, Taipei, Taiwan